CLINICAL TRIAL: NCT07398300
Title: Dynamic Whole-Body FDG and H₂¹⁵O PET-CT to Assess Insulin-Mediated Glucose Uptake and Organ Perfusion During GIP and GLP-1 Infusion in Healthy Individuals and Patients With Type 2 Diabetes
Brief Title: Insulin-Mediated Glucose Uptake and Organ Perfusion Assessed by Total-Body PET During GIP and GLP-1 Infusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mathilde Borring Brogaard, Doctor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H-25055805
Record Dates: First submitted 2026-01-28; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Healhty
Keywords: IncretinPET
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucagon-Like Peptide 1; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Two randomized crossover studies: Sub-study 1 uses a 3-period crossover (GIP, GLP-1, placebo) in healthy individuals; Sub-study 2 uses a 2-period crossover (GIP, GLP-1) in healthy individuals and participants with type 2 diabetes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GIP infusion (Experimental)
  Interventions: Drug: GIP
- GLP-1 infusion (Experimental)
  Interventions: Drug: GLP-1
- Saline Placebo (Experimental)
  Interventions: Other: Saline (0.9% Sodium Chloride)

INTERVENTIONS:
Drug: GIP — Intravenous infusion of glucose-dependent insulinotropic polypeptide (GIP) consisting of a priming dose of 18 pmol/kg/min for 10 minutes followed by a steady-state infusion of 6 pmol/kg/min during a hyperglycemic clamp. Used to stimulate endogenous insulin secretion and mimic postprandial physiology
  Arms: GIP infusion
Drug: GLP-1 — Intravenous infusion of glucagon-like peptide-1 (GLP-1) consisting of a priming dose of 4.5 pmol/kg/min for 10 minutes followed by a steady-state infusion of 1.5 pmol/kg/min during a hyperglycemic clamp. Used to stimulate endogenous insulin secretion and mimic postprandial physiology.
  Arms: GLP-1 infusion
Other: Saline (0.9% Sodium Chloride) — Intravenous infusion of isotonic saline administered as placebo. In sub-study 1, saline serves as a control condition; in sub-study 2, saline is infused for 15 minutes prior to hormone infusion.
  Arms: Saline Placebo

SUMMARY:
This study investigates how the naturally occurring gut hormones GIP and GLP-1 influence whole-body glucose uptake and organ perfusion in humans. Using a state-of-the-art total-body PET-CT scanner, the study measures dynamic uptake of the glucose analogue 18F-FDG and blood flow using H₂¹⁵O across multiple organs during controlled elevations of plasma glucose and endogenous insulin secretion.

The project consists of two sub-studies. Sub-study 1 includes healthy individuals who undergo three experimental visits with infusions of GIP, GLP-1, or saline (placebo) during a hyperglycemic clamp followed by FDG PET-CT scanning.

Sub-study 2 includes healthy individuals and participants with type 2 diabetes who undergo two experimental visits with saline followed by either GIP or GLP-1 during a hyperglycemic clamp, combined with repeated H₂¹⁵O PET-CT measurements of perfusion.

The primary aims are to quantify insulin-mediated skeletal muscle glucose uptake (sub-study 1) and skeletal muscle perfusion (sub-study 2). Secondary aims include assessment of glucose uptake and perfusion across adipose tissue, liver, and additional organs. The results will provide novel physiological insight into postprandial glucose metabolism and serve as reference data for future whole-body PET research.

ELIGIBILITY:
Sub-study 1 (Healthy individuals):

* Age 23-50 years
* BMI 20.0-26.9 kg/m²
* HbA1c < 42 mmol/mol
* Able to provide informed consent

Sub-study 2 - Participants with Type 2 Diabetes:

* Age 23-60 years
* Diagnosed with type 2 diabetes for ≥3 months
* HbA1c > 53 mmol/mol
* Treatment with metformin only
* Able to provide informed consent

Sub-study 2 - Healthy control participants:

* Age 23-64 years
* HbA1c < 42 mmol/mol
* Able to provide informed consent

Exclusion Criteria (applies to all participants unless otherwise specified):

* Anaemia (haemoglobin below normal range)
* ALT > 2× upper normal limit or any known hepatobiliary or gastrointestinal disorder
* Kidney disease (creatinine above normal range)
* Previous gastric or intestinal resection (except appendectomy or cholecystectomy) or major abdominal surgery (including bariatric surgery)
* For Sub-study 1: Type 1 or type 2 diabetes or HbA1c ≥ 42 mmol/mol
* Use of glucose-lowering medications other than metformin (Sub-study 2 only)
* Chronic obstructive pulmonary disease (Sub-study 2 only)
* Regular tobacco smoking or use of nicotine-containing products
* Claustrophobia
* Pregnancy, breastfeeding, or intention to become pregnant during the study period
* Initiation of special diets, major lifestyle changes, or weight loss > 5% within 3 months prior to or during the study
* Any medication or physical/psychological condition that may interfere with participation (per investigator judgement)
* Inability to speak or read Danish

Ages: 23 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-03-12 (Estimated); Primary Completion 2027-03-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Metabolic Rate of FDG | 75 minuts
  MRFDG quantified using dynamic total-body 18F-FDG PET with 3-compartment kinetic modelling during infusion of GIP, GLP-1, or placebo.

SECONDARY OUTCOMES:
Perfusion of skeletal muscle | 75 min

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital - Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No